CLINICAL TRIAL: NCT05621590
Title: MLC901 in Hypoxic-ischemic Brain Injury Patients; A Double-blind, Randomized Placebo-controlled Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Amini Harandi, associate professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.SBMU.RETECH.REC.1400.510
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Hypoxic Ischaemic Encephalopathy Due to Cardiac Arrest
MeSH Terms: interventions — Neuroaid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mlc-901 group (Experimental)
  Interventions: Drug: MLC 901
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MLC 901 — MLC901, also known as NeuroAiDII, is a capsule form of drug which should be taken orally and combines nine herbal components
  Other Names: Nueroaid II
  Arms: mlc-901 group
Drug: Placebo — placebo capsules filled with stevia sweetened powder
  Arms: placebo group

SUMMARY:
In a randomized, placebo-controlled trial, 35 patients with HIBI were randomly designated to receive either MLC901 or placebo capsules over six months.

We evaluated patients in two groups by modified Rankin Scale (mRS) and Glasgow outcome scale (GOS) to examine their state of disability and recovery

ELIGIBILITY:
Inclusion Criteria:

* an initial cardiac arrest leading to coma, successful return of spontaneous circulation, and persistent coma after the return of spontaneous circulation.

Exclusion Criteria:

* pregnancy, cardiogenic shock (systolic blood pressure less than 90 mm Hg despite epinephrine infusion), possible causes of coma other than cardiac arrest (drug overdose, head trauma, or cerebrovascular accident), an underlying background of known acute or chronic disease including renal failure, liver or pulmonary disorders, previous stroke, dementia, and brain injury.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
neurofunctional outcome using Glasgow Outcome Scale (GOS) | 6 months
neurofunctional outcome using modified Rankin Scale (mRS) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Beheshti University of Medical Sciences, Shohada Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pakdaman H, Amini Harandi A, Gharagozli K, Abbasi M, Ghaffarpour M, Ashrafi F, Delavar Kasmaei H, Amini Harandi A. MLC601 in vascular dementia: an efficacy and safety pilot study. Neuropsychiatr Dis Treat. 2017 Oct 5;13:2551-2557. doi: 10.2147/NDT.S145047. eCollection 2017. PMID 29042785